CLINICAL TRIAL: NCT07345780
Title: This Study is a Single-arm, Multicenter Investigator-Initiated Trial (IIT) Clinical Study. The Primary Objective is to Evaluate the Safety, Pharmacokinetic Characteristics, and Preliminary Efficacy of CAR-T Cells in Subjects With Relapsed/Refractory (r/r) CD7-positive Hematological Malignancies. The Study Plans to Enroll 20 Subjects, With the Actual Sample Size to be Determined Based on Real-world Occurrence.
Brief Title: Clinical Study on the Safety and Efficacy of CD7-Targeted Chimeric Antigen Receptor (CAR) Gene-Modified T Cells for the Treatment of CD7-Positive Hematological Malignancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-F
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: CD7-Positive Hematological Malignancies
MeSH Terms: interventions — Automobiles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:Experimental group (Experimental)
  Interventions: Drug: CD7-Targeted Chimeric Antigen Receptor (CAR) Gene-Modified T Cells for the Treatment of CD7-Positive Hematological Malignancies

INTERVENTIONS:
Drug: CD7-Targeted Chimeric Antigen Receptor (CAR) Gene-Modified T Cells for the Treatment of CD7-Positive Hematological Malignancies — CD7-Targeted Chimeric Antigen Receptor (CAR) Gene-Modified T Cells for the Treatment of CD7-Positive Hematological Malignancies

SUMMARY:
This study is a single-arm, multicenter Investigator-Initiated Trial (IIT) clinical study. The primary objective is to evaluate the safety, pharmacokinetic characteristics, and preliminary efficacy of CAR-T cells in subjects with relapsed/refractory (r/r) CD7-positive hematological malignancies. The study plans to enroll 20 subjects, with the actual sample size to be determined based on real-world occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their guardians understand and voluntarily sign the informed consent form, and are expected to complete the follow-up examinations and treatments required by the study protocol.

Aged 18-85 years (inclusive), gender not restricted. Subjects diagnosed according to WHO 2016 criteria with relapsed/refractory acute T-lymphoblastic leukemia/lymphoma (including early T-precursor lymphoblastic leukemia) who have failed standard treatment or lack effective treatment options, meeting any of the following criteria:a) Relapsed: Previously received at least two treatment regimens and achieved complete remission followed by confirmed disease recurrence, or achieved complete remission after stem cell transplantation followed by disease recurrence.b) Refractory: Previously received at least two treatment regimens and failed to achieve CR (for leukemia patients) or PR (for lymphoma patients) after the last treatment, or failed to achieve remission or experienced disease progression after stem cell transplantation.

Diagnosed with AML according to the 2016 WHO classification and meeting the diagnostic criteria for relapsed and refractory AML in the Chinese Guidelines for Diagnosis and Treatment of Relapsed/Refractory Acute Myeloid Leukemia (2017 Edition):a) Diagnostic criteria for relapsed AML: Reappearance of leukemic cells in peripheral blood after complete remission (CR), or >5% blasts in bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy), or extramedullary leukemic cell infiltration.b) Diagnostic criteria for refractory AML: Newly diagnosed cases failing to respond to standard treatment after 2 courses; Relapse within 12 months after CR following consolidation/intensification therapy; Relapse after 12 months but unresponsive to conventional chemotherapy; Two or more relapses; Persistent extramedullary leukemia.

Hematolymphoid malignancies confirmed by flow cytometry in bone marrow examination and/or by pathological immunohistochemistry in tumor tissue as CD7-positive at screening, with tumor positivity rate ≥70%.

Patients who have not received allogeneic hematopoietic stem cell transplantation (allo-HSCT) must have the ability to donate autologous mononuclear cells (hereinafter referred to as apheresis) or peripheral blood for CAR-T cell manufacturing. Peripheral blood smear at screening should show <30% tumor cells. For patients who have received allo-HSCT requiring autologous blood collection, peripheral blood smear at screening should also show <30% tumor cells; there is no such restriction if collecting donor blood.

Patients have recovered from the toxicity of previous treatments, i.e., CTCAE toxicity grade <2 (unless the abnormality is tumor-related or judged by the investigator to be stable with minimal impact on safety or efficacy).

ECOG performance status score 0-2 and life expectancy >3 months.

Appropriate organ function:

Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3×upper limit of normal (ULN). For ALT and AST abnormalities judged by the investigator to be disease-related (e.g., liver infiltration or biliary obstruction), the limit may be extended to ≤5×ULN.

Total bilirubin ≤1.5×ULN. Serum creatinine ≤1.5×ULN, or creatinine clearance ≥60 mL/min. Hemoglobin ≥60 g/L or maintained at this level after transfusion. Room air oxygen saturation ≥92%. Left ventricular ejection fraction (LVEF) ≥45%. Patients failing to meet any of the above criteria will not be enrolled as subjects.

Exclusion Criteria:

* History of malignancy other than T-cell hematological malignancies within 5 years prior to screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical treatment, and ductal carcinoma in situ of the breast after radical treatment.

Patients with clinically symptomatic central nervous system leukemia. Positive for hepatitis B surface antigen (HBsAg); positive for hepatitis B core antibody (HBcAb) with HBV DNA titer outside the normal reference range; positive for hepatitis C virus (HCV) antibody; positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA; positive for syphilis.

History of severe allergies [severe allergy defined as grade 2 or higher allergic reaction with any of the following clinical manifestations: airway obstruction (rhinorrhea, cough, wheezing, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory or cardiac arrest] or known hypersensitivity to any active ingredients, excipients, murine products, or xenogeneic proteins contained in this study (including lymphodepletion regimens).

Severe heart disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (defined as: blood pressure not controlled despite ≥3 antihypertensive drugs (including diuretics) at maximum tolerated doses for >1 month after lifestyle modification, or requiring ≥4 antihypertensive drugs for effective control).

Unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney, or metabolic diseases requiring medical treatment.

Previous organ transplantation or planned organ transplantation (except hematopoietic stem cell transplantation).

Acute or chronic graft-versus-host disease (GVHD) of any grade occurring 2 weeks after discontinuation of immunosuppressive therapy.

Hematopoietic stem cell transplantation within 6 months prior to screening. Active autoimmune or inflammatory neurological diseases (e.g., Guillain-Barré syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).

Tumor emergencies requiring urgent treatment at screening or prior to infusion (e.g., spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome).

Uncontrolled bacterial, fungal, viral, or other infections requiring antibiotic treatment.

Major surgery (except diagnostic procedures and biopsies) within 4 weeks prior to lymphodepletion or planned major surgery during the study, or incompletely healed surgical wounds prior to enrollment.

Live virus vaccination within 4 weeks prior to screening. Severe mental illness. History of alcoholism or substance abuse. Pregnant or lactating women, and female subjects planning pregnancy within 2 years after cell infusion or male subjects whose partners plan pregnancy within 2 years after their cell infusion.

Patients with contraindications to any study procedures or other medical conditions that may put them at unacceptable risk according to investigator judgment and/or clinical standards.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time frame:1, 3,6,12,18, 24 months after tretment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China